CLINICAL TRIAL: NCT02175784
Title: Postmarketing Clinical Study of Ipragliflozin - Double-blind, Parallel-group Study in Combination With Insulin in Patients With Type 2 Diabetes Mellitus
Brief Title: A Study to Assess the Efficacy and Safety of Ipragliflozin in Combination With Insulin in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1941-CL-0131
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Blood glucose; insulin; ipragliflozin; SGLT2 inhibitor
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — ipragliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ipragliflozin group (Experimental): oral
  Interventions: Drug: ipragliflozin
- placebo group (Experimental): oral
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ipragliflozin — oral
  Other Names: ASP1941; Suglat
  Arms: ipragliflozin group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
The purpose of this study is to assess the efficacy (superiority to placebo) of ipragliflozin based on the changes in HbA1C, as well as its safety, in patients with type 2 diabetes mellitus in combination with an insulin preparation once daily for 16 weeks. The long-term (52 weeks) safety and the persistence of the efficacy will also be evaluated.

DETAILED DESCRIPTION:
This study consists of two parts. First part is a placebo-controlled multicenter, double-blind, parallel group study, in which subjects will receive ipragliflozin or placebo once daily in combination with an insulin preparation for 16 weeks. Second part is a multicenter, open-label period (36 weeks) with no placebo group. The dose of ipragliflozin can be doubled in combination with an insulin preparation during the second part.

ELIGIBILITY:
Inclusion Criteria:

* Subject has been diagnosed with type 2 diabetes mellitus for at least 12 weeks (84 days) at signing of informed consent.
* Subject takes constant dosage and administration of insulin preparation for more than 6 weeks (42 days)
* Subject has an HbA1C value between 7.5 and 10.0% at Visit 2 and the difference of HbA1C value within ± 1.0% between Visit 1 and Visit 2
* Subject has a body mass index (BMI) 20.0 - 45.0 kg/m2

Exclusion Criteria:

* Subject has type 1 diabetes mellitus
* Subject has proliferative diabetic retinopathy
* Subject has a history of clinically significant renal disease such as renovascular occlusive disease, nephrectomy and/or renal transplant
* Subject has a history of recurrent urinary tract infection (more than three times within before 24 weeks of obtaining informed consent)
* Subject has a symptomatic urinary tract infection or symptomatic genital infection
* Subject has chronic disease which requires the continuous use of adrenocortical steroids and immunosuppressant (oral medication, injection, or inhalation)
* Subject has a history of cerebral vascular attack, unstable angina, myocardial infarction, vascular intervention, and heart disease (NYHA Class III-IV) within 1 year (52 weeks) prior to Visit 1
* Subject has unstable psychiatric disorder
* Female subject who is currently pregnant or lactating, or who is possibly pregnant
* Male and pre-menopausal female subject who cannot use an appropriate contraception during the study
* Subject has severe infection, perioperative, or serious trauma
* Subject has drug addiction or alcohol abuse
* Subject has a history of malignant tumors (except for those who have not received treatment for malignant tumors for at least 5 years before informed consent acquisition and was not considered to have recurrence)
* Subject has a history of an allergy with ipragliflozin and/or similar drugs (study drugs possessing SGLT 2 inhibitory action)
* Subject has participated in another clinical study, post marketing study, or medical equipment study within 12 weeks (84 days) before providing written informed consent, or who is currently participating in any of those studies
* Subject is unable, unwilling to adhere to compliances such as hospital visits and dose instruction specified in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2014-03-31 (Actual); Primary Completion 2015-03-31 (Actual); Study Completion 2015-12-07 (Actual)

PRIMARY OUTCOMES:
Change in HbA1C from baseline | Baseline and Week 16

SECONDARY OUTCOMES:
Fasting plasma glucose | Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Leptin concentration | Baseline, Week 2, 4, 8, 12, 16, 24, 36, 52
Fructosamine concentration | Baseline, Week 2, 4, 8, 12, 16, 24, 36, 52
Adiponectin concentration | Baseline, Week 2, 4, 8, 12, 16, 24, 36, 52
Body weight | Baseline, Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52
Waist circumference | Baseline, Week 16, 24, 52
Blood glucose values of self monitoring | Baseline, Week 8, 16, 24, 52
  written in a diary
Safety assessed by the adverse events, vital signs. and laboratory tests | Up to 52 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Kashiwagi A, Shestakova MV, Ito Y, Noguchi M, Wilpshaar W, Yoshida S, Wilding JPH. Safety of Ipragliflozin in Patients with Type 2 Diabetes Mellitus: Pooled Analysis of Phase II/III/IV Clinical Trials. Diabetes Ther. 2019 Dec;10(6):2201-2217. doi: 10.1007/s13300-019-00699-8. Epub 2019 Oct 12. PMID 31606880
- [Derived] Ishihara H, Yamaguchi S, Nakao I, Asahina S, Sakatani T. Efficacy and safety of ipragliflozin as add-on therapy to insulin in Japanese patients with type 2 diabetes mellitus (IOLITE): a 36-week, open-label extension of a 16-week, randomized, placebo-controlled, double-blind study. Diabetol Int. 2018 Jul 16;10(1):37-50. doi: 10.1007/s13340-018-0359-x. eCollection 2019 Jan. PMID 30800562
- See also: Link to results on Astellas Clinical Study Results website — https://www.astellasclinicalstudyresults.com/hcp/study.aspx?ID=171